CLINICAL TRIAL: NCT03932370
Title: Flexible Ureteroscopy Versus Mini-Percutaneous Nephrolithotomy for Treatment of Renal Stones 2 Cm or Less; A Randomised, Comparative Study.
Brief Title: Flexible Ureteroscopy Versus Mini-Percutaneous Nephrolithotomy for Treatment of Renal Stones
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Esam Saad Mohamed Darwish, assistant lecturer of urology, Assiut University
Other Study IDs: NCT03932370
Record Dates: First submitted 2019-04-27; First posted 2019-04-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Stone;Renal
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- f-URS
  Interventions: Procedure: Flexible ureteroscopy
- mini-PCNL
  Interventions: Procedure: mini-Percutaneus nephrolithotomy

INTERVENTIONS:
Procedure: Flexible ureteroscopy — The procedure will be performed in an endourology room where a radiolucent operative table together with a C-arm, a video-camera unit and a Laser device are available. Irrigation fluids include normal saline and/or sterile water.
  Other Names: RIRS; f.URS; Retrograde Intrarenal Surgery
  Groups: f-URS
Procedure: mini-Percutaneus nephrolithotomy — The procedure is done in the prone position under fluoroscopy guidance with a semi-rigid 12Fr. Nephroscope
  Other Names: Mini-perc; Mini-PCNL; m.PCNL
  Groups: mini-PCNL

SUMMARY:
Management of nephrolithiasis is evolving rapidly, and various minimally-invasive urological procedures are currently available for treating patients with renal stones, including extracorporeal shockwave lithotripsy (ESWL), flexible ureteroscopy (f-URS) and miniaturised percutaneous nephrolithotomy (mini-PCNL).

Despite being the only truly-non-invasive, outpatient procedure, stone-free rates (SFRs) of ESWL are lower than both mini-PCNL and f-URS. Furthermore, ESWL has several limitations, such as pregnancy; uncorrected coagulopathy;aortic aneurism; severe obesity; large stone burdens (>2cm); stones with high densities (>970/1000 Hounsfield units); ESWL-resistant stone compositions; lower calyceal stones with unfavourable anatomical criteria; and stones in calyceal diverticula; Morbidities of the conventional PCNL are significantly minimised by using less access diameters in PCNL while providing comparable SFRs. Additionally, Mini and Micro PCNL result in shorter hospital stay and higher tubeless rates compared to conventional PCNL.

Flexible ureteroscopy has been increasingly used as a primary modality for treatment of renal stones with significantly lower complication rates than PCNL and mini-PCNL in terms of less bleeding and transfusion rates, shorter hospital stay and less postoperative pain. Additionally, f-URS is the only treatment modality of nephrolithiasis that can be safely and effectively used in patients with bleeding tendency, as well as pregnant women; moreover, its outcomes are not affected by obesity. Nevertheless, its poor durability and high costs remain major limitations for f-URS, especially in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Age above than 15 years
* Renal stone(s) with total burden of 2 cm or less
* Signature on written, informed consents with the details of this study requirements.
* Inappropriateness or failure of ESWL (examples of ESWL inappropriateness: patient preference; distal obstruction; contraindications of ESWL)

Exclusion Criteria:

* Uncorrectable bleeding diathesis
* Current pregnancy

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: no specific criteria
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
initial stone clearance | 24 hours after the operation
  Number of participants who has been totally cleared of stones as measured by KUB and ultrasound
final stone clearance | 90 days after the operation
  Number of participants who has been totally cleared of stones as measured by non-contrast CT

SECONDARY OUTCOMES:
Operative time | Within 24 hours
  time passed during the operation
Hospital stay | Within a week from the operation
  Number of days the patient has been hospitalised
Haemoglobin drop | within 24 hours
  The percentage of haemoglobin drop before and after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Urology and Nephrology Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No